CLINICAL TRIAL: NCT00768209
Title: A Phase I, Open Label, Single-Dose Study to Evaluate the Pharmacokinetics of VI-0521 in Subjects With Hepatic Impairment and In Healthy Control Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics of VI-0521 in Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Collaborators: Covance (Industry); Sentrx (Industry)
Responsible Party: Wesley Day, VP Clinical, Vivus, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OB-105
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Hepatic Impairment
Keywords: Pharmacokinetics
MeSH Terms: interventions — Qsymia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment A (Experimental)
  Interventions: Drug: Phentermine and Topiramate

INTERVENTIONS:
Drug: Phentermine and Topiramate — Each subject will be dosed with a single oral dose of VI-0521 (PHEN/TPM 15/92 mg).

SUMMARY:
This study is designed to determine the effects of a single dose of the study medication in subjects with and without hepatic impairment. 18 to 24 subjects will participate by having multiple blood draws taken to measure the level of study medication in their blood over time.

DETAILED DESCRIPTION:
This study will look at the effect of a single does of study medication in three groups. Each group will have 6 - 8 subjects with similar levels of hepatic impairment. Group 1 will have normal hepatic function. Groups 2 and 3 will be made up of subjects with mild to moderate hepatic impairment. Subjects will have blood taken at specific intervals to measure study medication levels. Subject participation will last approximately 7 to 9 days.

ELIGIBILITY:
Inclusion Criteria:

A total of 18 to 24 subjects will be studied in 3 groups of 6-8 subjects per group. Group 1 will consist of 6-8 males or females with normal hepatic function, 18 to 65 years of age inclusive. Groups 2-3 will consist of 6-8 males or females per group with varying degree of stable hepatic impairment.

Exclusion Criteria:

Any Subject meeting the following criteria must be excluded from the trial:

1. Known history of clinically significant arrhythmias.
2. Acute illness, especially any infection, within 2 weeks of dosing.
3. History or presence of:

   * Alcoholism or drug abuse within the past 2 years.
   * Hypersensitivity or idiosyncratic reaction to compounds related to the study drug or related compounds.
4. Any History of Bipolar disorder or psychosis, history of psychiatric hospitalization, greater than one lifetime episode of major depression.
5. Blood donation or significant blood loss within 56 days prior to Day 1.
6. Plasma donation within 7 days prior to Day 1.
7. Any subject who has participated in a previous clinical trial with VI-0521.
8. Any subject who received an investigational drug within 30 days prior to dosing in this study.
9. Any history of glaucoma, increased intraocular pressure, or medications to treat increased intraocular pressure.
10. Serum creatinine > 1.5 for male subjects, and >1.4 for female subjects.
11. History of kidney stones in the last 6 months
12. Female subjects, who may be pregnant, or are lactating.
13. Use of any drug that is known to have clinical significance in inhibiting or inducing liver enzymes involved in drug metabolism.
14. Use of tobacco or nicotine products within last 6 months unless subject is hepatically-impaired.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Shiyin Yee, PhD, Study Director — VIVUS LLC
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida